CLINICAL TRIAL: NCT05754034
Title: Building Respiratory Support in East Africa Through High Flow Versus Standard Flow Oxygen Evaluation
Acronym: BREATHE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, Elisabeth Riviello, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P001102; 222165/Z/20/Z (Other Grant/Funding Number: Wellcome Trust (WT))
Record Dates: First submitted 2023-02-07; First posted 2023-03-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Hypoxemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High flow oxygen (Experimental): Heated and humidified oxygen delivered via high flow oxygen device through nasal cannula, up to 60 liters per minute of flow.
  Interventions: Device: High flow oxygen
- Standard flow oxygen (Active Comparator): Oxygen delivered via standard oxygen devices at standard flows up to 15 liters per minute: nasal cannula, face mask, or nonrebreather mask.
  Interventions: Other: Standard flow oxygen

INTERVENTIONS:
Device: High flow oxygen — humidified and heated oxygen delivered at high flow rates via nasal cannula, with protocol to target SpO2 90-94%
  Arms: High flow oxygen
Other: Standard flow oxygen — oxygen delivered at standard flow rates via nasal cannula, facemask, or nonrebreather mask, with protocol to target SpO2 90-94%
  Arms: Standard flow oxygen

SUMMARY:
Acute hypoxemia is common and deadly in resource variable settings. While studies in high income countries (HICs) have indicated a possible benefit to high flow oxygen as compared with standard flow oxygen, rigorous studies in low or lower middle income countries (LMICs) have not been performed. Studies in sepsis have demonstrated that interventions that improve outcomes in one context may actually be neutral or harmful in a different context.

The goal of this study is to test whether high flow oxygen results in better outcomes for hypoxemic adult patients, as compared with standard flow oxygen, in five LMIC hospitals. The main questions it aims to answer are:

1. For hypoxemic adults in these LMIC study settings, does high flow oxygen or standard flow oxygen result in lower mortality?
2. What are the facilitators and barriers to using high flow oxygen in these settings?
3. Does high flow or standard flow oxygen use more oxygen?

Participants will be randomized to receive either high flow oxygen through a large nasal cannula, or to receive standard flow oxygen, through nasal cannulas, face masks, or non-rebreather masks. Researchers will compare the outcomes for the two groups, to see if one group of patients has better outcomes than the other.

The study will also examine how much oxygen is used by the two patient groups, as well as other factors relevant to the feasibility of implementation of high flow oxygen in these sites.

ELIGIBILITY:
Inclusion Criteria:

* age>=18 years AND
* admitted to a study site hospital within the 24 hours prior to screening AND
* SpO2<90% at time of first assessment OR
* receiving oxygen at time of first assessment

Exclusion Criteria:

* imminent death (high clinical suspicion of death within 24 hours of admission)
* patient or caregiver refusal of study participation
* history of chronic respiratory failure (SpO2<90% or oxygen dependence for at least three months)
* anatomical factors precluding the use of nasal cannula
* intubation or non-invasive ventilation by the clinical team prior to screening for the trial
* known hypoxemia at transferring facility for >48 hours
* lack of availability of either SFO or HFO devices or supplies at the time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Day 90
  Death between randomization and end of hospitalization

SECONDARY OUTCOMES:
90-day mortality | Day 90
  Death between randomization and 90 days
90-day functional status | Day 90
  Functional status 90 days after randomization, as measured by the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
Need for mechanical ventilation | Day 90
  Met objective criteria for need to escalate respiratory therapy to NIV or invasive ventilation, or escalated to NIV or mechanical ventilation
Days requiring oxygen | Day 90
  Days requiring oxygen from randomization to end of hospitalization
Hospital length of stay | Day 90
  Days from randomization to hospital discharge or death
ICU length of stay | Day 90
  Total days in the ICU during hospitalization
Time to meeting criteria for need for escalation to either NIV or invasive ventilation | Day 90
  Time to meeting objective clinical criteria for escalation to non-invasive ventilation or invasive ventilation
Time to escalation to either NIV or invasive ventilation | Day 90
  Time to escalation to non-invasive ventilation or invasive ventilation

OTHER OUTCOMES:
Oxygen consumption | Day 90
  Total oxygen consumed during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Riviello, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- Kenya (2):
  - AIC Kijabe Hospital, Kijabe
  - Nakuru Level V Hospital, Nakuru
- Queen Elizabeth Central Hospital, Blantyre, Malawi
- Rwanda (2):
  - The University Teaching Hospital of Butare (CHUB), Huye
  - The University Teaching Hospital of Kigali (CHUK), Kigali

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers for the trial overall. IPD is owned and managed by each of the sites for the trial, in accordance with the data protection requirements of each country where the sites are located. Individual sites may decide to share their own IPD with other researchers.